CLINICAL TRIAL: NCT04137016
Title: Pilot Study to Assess the Impact of a Mobile Health Application (App) on Clinical Outcomes and Satisfaction of Older HIV-Infected Patients, as an Emerging Tool for Care, Education and Prevention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APP-Age
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-10

CONDITIONS: HIV-1 Infection
Keywords: APP, old
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-subjects with APP (Experimental): HIV-infected patients using the App + standard clinical management (SCM)
  Interventions: Other: Mobile application
- Control group (No Intervention): HIV-infected patients, who only receive Standard Clinical Management (without the App)

INTERVENTIONS:
Other: Mobile application
  Arms: HIV-subjects with APP

SUMMARY:
In recent years, HIV care has been reframed by the concepts of the HIV care and prevention. The success of these strategies will depend on integrated prevention and care system and sustained behavioral modification. The HIV infection is a chronic disease and the improved survival in HIV patients favours the emergence of new long-term morbidities associated with treatment and/or the virus itself. In high-income countries, approximately 30% of all adults living with HIV are aged 50 years and over. In 2015, 50% of HIV-infected patients will be over 50 years of age. Health plans are a priority to prevent this accelerated and accentuated process.

The development of mobile devices such as smartphones and tablet computers has spurred rapid growth in the field of mobile health, the use of mobile-enabled applications that collect or deliver health care information and data. These applications offer the potential for dynamic engagement of patients and providers in health care and a new means of improving health outcomes. This technology could have profound application in the prevention or in the treatment of patients with chronic disease such as diabetes, obesity, HIV, etc, since these diseases are generating more health spending worldwide. The rapid growth in health has outpaced the needed to validate the clinical effectiveness of these applications. For this reason, we propose a study to assess the benefit of a specific App on the management of HIV-infected population aged 60 years or older It is a Randomized clinical trial, including 2 groups: 1) an experimental group comprising patients using the app + routine medical care and 2) a control group. The usability of the app and patient satisfaction were evaluated in the app group at weeks 24 and 48. Quality of life, adherence to treatment, and clinical parameters were compared in both groups at 48 weeks.

DETAILED DESCRIPTION:
Aging is the term used to describe the progressive loss of physical ability, changes in appearance, and/or decrease in mental agility that we experience over time. This process advances at different rates as a consequence of genetic and environmental factors.

Aging of the population can be considered a success of public health policies and socioeconomic development, although it also constitutes a challenge for society, which must adapt in order to improve the health and functional capacity of the elderly, as well as their social participation and their safety.

However, a recent major study on health and aging warned that the burden of chronic disease will considerably affect quality of life in aging patients.

The increase in the average age worldwide makes chronic diseases and the consequent reduction in well-being a prominent global public health challenge. One of the greatest challenges for a national health system is to achieve sustained care of people with chronic health problems (both physical and psychological).

HIV infection is a chronic disease. However, the life expectancy of affected patients has increased considerably thanks to advances in antiretroviral treatment. In 2015, around 50% of HIV-infected patients were ≥50 years old. It is estimated that by 2030, around 70% of the HIV-infected population in the United States of America will be aged ≥50 years.

Growing evidence in the scientific literature suggests an increased prevalence of long-term comorbidities associated with antiretroviral treatment and the infection itself compared with noninfected controls of the same age. In addition, aging could manifest 10 years earlier with respect to the general population.

As a result, HIV infection is an increasingly complex chronic disease associated with numerous medical, psychological, and social problems that require the attention and experience of a wide range of health specialists.

Information and communications technologies are a strategic element in improving health and ensuring a quality, modern, and sustainable health system. The development of mobile devices such as smartphones and tablets has shown how mobile applications (apps) have revolutionized health care (medical apps). Information and communications technologies could prove very useful in the care of patients with chronic conditions, such as diabetes, obesity, and cardiovascular disease. They could also play a role in the prevention of comorbid conditions.

Considering that HIV infection is a chronic disease, our objective was to determine the usefulness of an app designed specifically for HIV-infected patients aged ≥60 years. To do so, we evaluated the usability of the application in this population and assessed changes in patient satisfaction with and quality of health care.

Since we did not know how familiarized this population was with mobile apps, we set a dual main objective: 1) before the clinical trial, participants completed an 8-item survey to determine their interest in medical apps and thus determine appropriate sections of interest; 2) to determine the usability of a specific app among HIV-infected patients aged ≥60 years by assessing, at week 24, the percentage of subjects randomized to the app who used the app on more than 10 different days after baseline. A final analysis was performed at week 48 to determine usability at the end of the study.

The secondary objectives were as follows: 1) to identify the most frequently used items in the app by comparing the items used with those that the patients mentioned in a survey at week 48; 2) to compare the number of visits to the HIV Unit in each group (app and controls); 3) to compare patient satisfaction in the app group by means of an ad hoc test ranging from 1 (worst) to 5 (best) between baseline and week 48; 4) to compare the groups by assessing adherence (SERAD), quality of life (MOS), and a series of clinical parameters at week 48.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients (≥60 years).
* Patients in antiretroviral treatment
* Patients who have and are used to a smartphone
* Patient who agree to participate in the study and signed informed consent

Exclusion Criteria:

- Patients with conditions that hampered understanding and use of mobile applications

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
The number of clinical events or comorbidities between the 2 groups | from baseline to week 48
change in bone mineral density Prevention | from baseline to week 48
  (BMD, lumbar and hip T-scores and Z-scores) measured by DXA scan.

SECONDARY OUTCOMES:
To compare patient satisfaction in the app group | Since baseline to week 48
  compare patient satisfaction in the app group by means of an ad hoc test ranging from 1 (worst) to 5 (best) between baseline and week 48
Usability of App | Since baseline to week 48
  • Assessing, at week 24, the percentage of subjects randomized to the app who used the app on more than 10 different days after baseline. A final analysis was performed at week 48 to determine usability at the end of the study.app on more than 10 different days after baseline. A final analysis was performed at week 48 to determine usability at the end of the study.
Identify the most frequently used items in the app | From baseline to week 48
  comparing the items used with those that the patients mentioned in a survey at week 48. We use a linkert Scale: minimum and maximum values: 1 low satisfied-5 higly satisfied
Quality of life (Global, physical, mental and social) | From baseline to Week 48
  compare the groups by assessing quality of life (Medical Outcomes Study-HIV Health Survey) with a questionnaire. 4 qualitative categories ( Global, physical, mental and social).: minimum and maximum values: very poor qualitiy of life; poor quality of life; good quality of life; very good quality of life.
adherence | From baseline to Week 48
  compare the groups by assessing quality of life (SERAD test)
Changes in FRAX equation. | From baseline to week48

OTHER OUTCOMES:
Changes in blood pressure, | From baseline to week48
Changes in glycemia | From baseline to week48
Changes in weight | The number of clinical visits at the HIV unit, and hospitalizations.
Changes in exercise | From baseline to week48
Changes in smoking habit | From baseline to week48
The number and severity of antiretroviral-related adverse events | From baseline to week48
The number of clinical visits at the HIV unit, and hospitalizations. | From baseline to week48

CONTACTS AND LOCATIONS:
Overall Officials: EUGÈNIA NEGREDO, PhD, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain